CLINICAL TRIAL: NCT04124419
Title: Baseline Controlled Study to Evaluate the Safety and Efficacy of Combined EMS and RF Treatments for Non-Invasive Circumference Reduction and Skin Tightening
Brief Title: Safety and Efficacy of Combined EMS and RF Treatments
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: InMode MD Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DO608715A
Record Dates: First submitted 2019-08-06; First posted 2019-10-11 (Actual); Last update posted 2021-08-25 (Actual); Status verified 2021-02

CONDITIONS: Non-invasive Circumference Reduction
MeSH Terms: interventions — Therapeutics

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Treatment Arm (Experimental): Eligible subjects will receive up to 3 treatments (2-week interval) with the Evolve device utilizing the Ti10 and Tone applicators according to the study protocol.
  Interventions: Device: Treatment with Evolve System

INTERVENTIONS:
Device: Treatment with Evolve System — EMS and RF Treatment

SUMMARY:
The objective of this trial is to evaluate the safety and efficacy of the Evolve device utilizing the Ti10 and Tone applicators for abdominal non-invasive circumference reduction and skin tightening

ELIGIBILITY:
Inclusion Criteria:

* - Signed informed consent to participate in the study.
* Female and male subjects,18 - 65 years of age at the time of enrolment
* BMI≤ 30
* If female, not pregnant, lactating and must be either post-menopausal, surgically sterilized, or using a medically acceptable form of birth control at least 3 months prior to enrolment (i.e., oral contraceptives, contraceptive implant, barrier methods with spermicide or abstinence).
* In addition, negative urine pregnancy test as tested before each treatment and at the last visit for women with childbearing potential (e.g. not menopause).
* General good health confirmed by medical history and skin examination of the treated area.
* Willing to have photographs and images taken of the treated areas to be used de-identified in evaluations, publications and presentations.
* The patients should be willing to comply with the study procedure and schedule, including the follow up visit, and will refrain from using any other aesthetic treatment methods for the last 6 months and during the entire study period.

Exclusion Criteria:

* - Pacemaker or internal defibrillator, or any other metallic or electronic implant anywhere in the body.
* Permanent implant in the treated area such as metal plates, screws and metal piercing, silicone implants or an injected chemical substance, unless deep enough in the periosteal plane.
* Intra-dermal or superficial sub-dermal areas that have been injected with HA/collagen/fat injections or other augmentation methods with bio-material during last 6 months.
* Current or history of skin cancer, or current condition of any other type of cancer, or pre-malignant moles.
* Severe concurrent conditions, such as cardiac disorders, sensory disturbances, epilepsy, uncontrolled hypertension, and liver or kidney diseases.
* Pregnancy and nursing.
* Impaired immune system due to immunosuppressive diseases such as AIDS and HIV, autoimmune disorders or use of immunosuppressive medications.
* Patients with history of diseases stimulated by heat, such as recurrent Herpes Simplex in the treatment area, may be treated only following a prophylactic regimen.
* Poorly controlled endocrine disorders, such as diabetes or thyroid dysfunction and hormonal virilization.
* Any active condition in the treatment area, such as sores, psoriasis, eczema, and rash.
* History of skin disorders, keloids, abnormal wound healing, as well as very dry and fragile skin.
* History of bleeding coagulopathies, or use of anticoagulants in the last 10 days.
* Any surgical procedure in the treatment area within the last 6 months or before complete healing.
* Having received treatment with light, laser, RF, or other devices in the treated area within 3 months, or before complete healing.
* Use of Isotretinoin (Accutane®) within 6 months prior to treatment.
* As per the practitioner's discretion, refrain from treating any condition which might make it unsafe for the patient.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2019-07-19 (Actual); Primary Completion 2021-05-19 (Actual); Study Completion 2021-05-19 (Actual)

PRIMARY OUTCOMES:
Change in circumference reduction | 1 month, 3 month, 6 months
  statistical difference in circumference reduction between Control (baseline measurement) and three points of follow-up measurement: 4 weeks (1Month) 12 weeks (3Month) and 24 weeks (6 months) following the last Tx session.
Change in skin appearance | 1 month, 3 month, 6 months
  Improvement in skin appearance comparing pre and at 1, 3 months and 6 months post last treatment photographs (as assessed by blinded investigators):
  Success is defined by correct identification of the pre and post-treatment photos as demonstrated in at least 70% or greater of patients completed the treatment at 1 month, 3 months, and 6 months post-treatment.
Change in abdomen area appearance assessed by 3D Photographic analysis | 1 month, 3 month, 6 months
  3D Photographic analysis will be conducted using QuantifiCare System at follow up visits and compared to the baseline.
Change in abdomen area appearance assessed by Investigator | 1 month, 3 month, 6 months
  - Investigator assessment of the skin appearance comparing pre and post treatment using 0 - 4 -points Likert scale at follow up visits: 4 = Significantly marked improvement; 3 = Marked improvement; 2 = Moderate improvement; 1 = Slight improvement; 0 = No difference

SECONDARY OUTCOMES:
Subject Improvement assessment | 1 Month, 3 Months, 6 Months
  Improvement assessment will be performed independently by the subject himself using 4 points Likert scale questionnaire (Global Aesthetic Improvement Scale), as follows:
  4 = Significantly marked improvement; 3 = Marked improvement; 2 = Moderate improvement; 1 = Slight improvement; 0 = No difference.
Subject satisfaction assessment | 1 month, 3 months, 6 months
  Subject assessment of satisfaction will be filled out by subjects using a 5-points Likert scale, as follows:
  +2 = Very satisfied; +1 = Satisfied; 0 = Indifferent; -1 = Disappointed; -2 = Very disappointed.
Subject assessment of comfort | 1 month, 3 months, 6 months
  Subject assessment of comfort will be filled out by subjects using a 5-point Likert scale, as follows:
  +2 = Very comfortable; +1 = Comfortable; 0 = Indifferent; -1 = uncomfortable; -2 = Pain.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Avance Plastic Surgery Institute, Reno, Nevada
  - BodySculpt, New York, New York